CLINICAL TRIAL: NCT01350791
Title: Evaluation of Effectiveness and Safety of PROMUS Element™ in Routine Clinical Practice; A Multicenter, PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: Evaluation of Effectiveness and Safety of PROMUS Element Stent (IRIS-ELEMENT )
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-04
Record Dates: First submitted 2011-04-22; First posted 2011-05-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Promus Element stent: Patients receiving Promus Element stents

SUMMARY:
This study is a non-randomized, prospective, open-label registry to compare the efficacy and safety of Promus Element stents versus first-generation drug-eluting stent (DES) in patients with coronary artery disease.

DETAILED DESCRIPTION:
The Element Stent platform features a proprietary Platinum Chromium Alloy, designed specifically for coronary stents. This alloy, coupled with a new stent architecture, is designed to enable thinner struts, increased flexibility and a lower profile while improving radial strength, recoil and visibility. In addition, the PROMUS Element Stent System incorporates the new Apex™ Dilatation Catheter technology, designed to enhance deliverability to complex lesions.

Currently, there have been limited data regarding comparison of PROMUS Element stent with first-generation DES in routine clinical practice. Therefore, we perform large-scale real-world registry of PROMUS Element stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Promus Element stents
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients with cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Coronary artery disease requiring drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 3001 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months post stenting procedure

SECONDARY OUTCOMES:
Death (all-cause and cardiac) | 30 days
Myocardial infarction | 30 days
Composite of death or MI | 30 days
Composite of cardiac death or MI | 30 days
Target Vessel Revascularization | 30 days
Target lesion revascularization | 30 days
Stent thrombosis | 30 days
Procedural success(defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization) | 3 days in average
  At discharge from the index hospitalization, participants will be followed for the duration of hospital stay, an expected average of 3 days.
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | yearly up to 5 years
Myocardial infarction | 6 months
Myocardial infarction | yearly up to 5 years
Composite of death or MI | 6 months
Composite of death or MI | yearly up to 5 years
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | yearly up to 5 years
Target Vessel Revascularization | 6 months
Target Vessel Revascularization | yearly up to 5 years
Target lesion revascularization | 6 months
Target lesion revascularization | yearly up to 5 years
Stent thrombosis | 6 months
Stent thrombosis | yearly up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center; Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea
Locations (1):
- 38 Centers, Seoul, South Korea